CLINICAL TRIAL: NCT00708396
Title: Tolerability And Efficacy Of High Dose Escitalopram In The Treatment Of Patients Suffering From Schizophrenia And Obsessive-Compulsive Disorder (OCD) - An Open Label Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: BeerYaakov Mental Health Center (Other Government)
Responsible Party: BeerYaakov Mental Health Center, BeerYaakov Mental Health Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Escitalopram -199CTIL
Record Dates: First submitted 2008-07-01; First posted 2008-07-02 (Estimated); Last update posted 2009-01-27 (Estimated); Status verified 2009-01

CONDITIONS: OCD; Schizophrenia
Keywords: Patients; suffer; from
MeSH Terms: conditions — Schizophrenia | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients (Experimental): Patients which diagnosed as OCD and schizophrenia
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — First week; 10mg/d of Escitalopram Weeks 2-5; 20mg/d of Escitalopram After 4 weeks of 20mg treatment (2-5 weeks of the study) - if partial/no response according to YBOCS score and clinical judgment, the dose will be increased up to 30mg for 4 weeks (weeks 6-9) and in case of partial/ non response the dose will be increased up to 40 mg until the completion of the study (weeks 10-13).

SUMMARY:
The purpose of the study is to evaluate tolerability and efficacy of escitalopram (Cipralex) treatment in doses beyond 20mg (20-40 mg/d) in patients with OCD and schizophrenia, non responsive or partially responsive to recommended doses (evaluation according to Y-BOCS).

An open label, prospective study. The study will include 20 patients recruited from the inpatient wards and from the outpatient clinic who have a DSM-IV diagnosis of schizophrenia or schizoaffective disorder and OCD.

Before entering the study all patients will be interviewed by 2 senior board certified psychiatrists in order to confirm the diagnosis of schizophrenia or schizoaffective disorder and OCD according to DSM-IV criteria.

After confirming the diagnosis of schizophrenia/schizoaffective disorder and OCD each patient will be evaluated by PANSS, Y-BOCS and GCI-S scales. Those patients who score above 12 points on the Y-BOCS will be eligible for the study.

Rating scales (PANSS, Y-BOCS, CGI-S, CGI-I) will be completed on a weekly basis during the whole 13 weeks period. In addition patients will be asked to report medication side effects and will also be clinically evaluated for side effects by the physician. Special attention will be paid to worsening of psychosis or OC symptoms. All patients whose mental status will deteriorate or those who cannot tolerate the drug will be dropped-out and intent to treat analysis will be made.

ELIGIBILITY:
Inclusion Criteria:

* All patients will be men and women over 18 years of age who meet DSM-IV criteria for schizophrenia/ schizoaffective disorder and OCD.
* Previous to entering the study all patients should be stabilized on antipsychotic medication for at least 3 months.
* Patients should score above 12 points on Yale Brown Obsessive Compulsive Scale (Y-BOCS) (Cut off point of Y-BOCS total score > or =7 is the common practice in similar studies) (Kayahan et al 2005).

Exclusion Criteria:

* All patients who are under antidepressant treatment (including SSRIs and clomipramine).
* In patients who were on clomipramine or SSRI in the past are included, at least 2 weeks must have been elapsed since stopping the medication.
* In case the patient has received an antidepressant which is not an SSRI or clomipramine, there will be a washout period of one week before entering the study.
* If the patient received a MAO-inhibitors there will be a washout period of at least 2 weeks except for fluoxetine for which a washout period of 5 weeks is required due to its long half-life.
* Known contraindication for the use of citalopram or escitalopram.
* Abnormal ECG findings at baseline
* Unable to understand and give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-07; Primary Completion 2010-07 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
1. Yale-Brown Obsessive Compulsive Scale (Y-BOCS) Symptom Checklist | on a weekly basis during the whole 13 weeks period
2. Positive and negative symptoms scale ( PANSS) | on a weekly basis during the whole 13 weeks period
3. The Clinical Global Impression scales (CGI) consist of two sub-scales: The Severity of illness (CGI-S) and the Global improvement (CGI-I). | on a weekly basis during the whole 13 weeks period
4. Blood lipids and blood glucose prior to escitalopram up-titration over 20mg/d and at last visit | on a weekly basis during the whole 13 weeks period
5. EKG and physical examination will be performed at baseline 6. AE checklist at every visit 7. Recent and concomitant medications at every visit | on a weekly basis during the whole 13 weeks period

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Octavio Stryjer, MD, Principal Investigator — Beer-Yaacov MHC
Locations (1):
- Beer-Yaacov MHC, Beer-Yaacov, Israel